CLINICAL TRIAL: NCT01106404
Title: RestoreSensor Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1651
Record Dates: First submitted 2010-04-02; First posted 2010-04-19 (Estimated); Results first posted 2012-08-01 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 6-week AdaptiveStim followed by 6-week manual programming (Other)
  Interventions: Device: RestoreSensor Neurostimulation System
- 6-week manual followed by 6-week AdaptiveStim programming (Other)
  Interventions: Device: RestoreSensor Neurostimulation System

INTERVENTIONS:
Device: RestoreSensor Neurostimulation System — Adjustments to stimulation settings are automatic when the AdaptiveStim feature of the device is turned "ON" and manual when the AdaptiveStim feature of the device is turned "OFF".

SUMMARY:
The purpose of the study is to gather clinical information on subjects' experiences with and without the use of the new feature of the RestoreSensor implantable neurostimulator (INS).

DETAILED DESCRIPTION:
This study is a multi-center, prospective, open-label, randomized, crossover study that is designed to gather clinical information on subjects' experiences with the use of the new feature of the RestoreSensor implantable neurostimulator. Current spinal cord stimulators for chronic intractable pain stimulate targeted nerves along the spine using electrical impulses. The stimulation interferes with the transmission of pain signals to the brain replacing painful sensations with a tingling sensation called paresthesia. Variation in the intensity of neurostimulation with body position is a challenge for some patients implanted with conventional spinal cord stimulation systems because positional changes may result in overstimulation or understimulation. Patients need to manually adjust their stimulation using the patient programmer to maintain their comfort level during position changes. The AdaptiveStim feature of the RestoreSensor neurostimulator was developed to address this challenge by improving pain relief and/or convenience relative to manual programming adjustments.

ELIGIBILITY:
Inclusion Criteria:

* Meets the indications as an appropriate surgical candidate (after successful SCS screening trial) for implant of a neurostimulation system for spinal cord stimulation (SCS) treatment of trunk and/or limb pain, per labeled indications
* 18 years of age or older
* Willing and able to attend visits and comply with the study protocol
* Capable of using the patient programmer and recharging the neurostimulator (INS), able to read and answer questionnaires in English, without assistance of a caregiver
* Males and non-pregnant females

Exclusion Criteria:

* Has had a prior implantable SCS neurostimulation system
* Currently enrolled, or plans to enroll in another investigational device or drug trial during the study
* Has unresolved legal issues related to their pain condition for which they would be receiving neurostimulation
* Requires cervical placement of leads.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Huntsville, Alabama
  - Oceanside, California
  - Edina, Minnesota
  - Las Vegas, Nevada
  - Voorhees Township, New Jersey
  - Eugene, Oregon
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Schultz DM, Webster L, Kosek P, Dar U, Tan Y, Sun M. Sensor-driven position-adaptive spinal cord stimulation for chronic pain. Pain Physician. 2012 Jan-Feb;15(1):1-12. PMID 22270733

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The sponsor activated 10 study centers after the study protocol was approved by FDA in March 2010. The overall recruitment for study subjects lasted less than 5 months, with the first enrollment on April 20, 2010, and last enrollment on September 3, 2010.
Pre-assignment Details: Among the 79 subjects enrolled into the study, there were 3 subjects discontinued prior to implantation. The reasons for discontinuations were withdrawal of consent (n = 2) and eligibility criteria not met (n = 1). A total of 76 subjects were implanted and randomized at 4 weeks post implant.
Groups:
- 6-week AdaptiveStim Followed by 6-week Manual Programming: Subjects received AdaptiveStim programming for 6 weeks, followed by manual programming for 6 weeks.
- 6-week Manual Followed by 6-week AdaptiveStim Programming: Subjects received manual programming for 6 weeks, followed by AdaptiveStim programming for 6 weeks.
Period: Period I (First 6 Weeks)
Arm/Group | 6-week AdaptiveStim Followed by 6-week Manual Programming | 6-week Manual Followed by 6-week AdaptiveStim Programming
Started | 36 | 40
Completed | 33 | 38
Not Completed | 3 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Period: Period II (Second 6 Weeks)
Arm/Group | 6-week AdaptiveStim Followed by 6-week Manual Programming | 6-week Manual Followed by 6-week AdaptiveStim Programming
Started | 33 | 38
Completed | 33 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6-week AdaptiveStim Followed by 6-week Manual Programming | 6-week Manual Followed by 6-week AdaptiveStim Programming | Total
Number analyzed (Participants) | 36 | 40 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 61
  >=65 years | 5 | 10 | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 52.5 (13.0) | 53.1 (14.1) | 52.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 27 | 45
  Male | 18 | 13 | 31
Region of Enrollment [Number; unit: participants]
  United States | 36 | 40 | 76
average Numeric Pain Rating Scale (NPRS) [Mean (Standard Deviation); unit: units on a scale] — NPRS is a 11-point scale with numbers from 0 to 10, with 0 meaning "No pain" and 10 meaning "Pain as bad as you can imagine." For average NPRS, study subjects were instructed to "Please rate your pain by indicating the number that best describes your pain on average in the last 24 hours."
  units on a scale | 6.26 (1.48) | 5.88 (2.15) | 6.06 (1.86)
worst Numeric Pain Rating Scale (NPRS) [Mean (Standard Deviation); unit: units on a scale] — NPRS is a 11-point scale with numbers from 0 to 10, with 0 meaning "No pain" and 10 meaning "Pain as bad as you can imagine." For worst NRPS, study subjects were instructed to "Please rate your pain by indicating the number that best describes your worst pain in the last 24 hours."
  units on a scale | 7.60 (1.15) | 7.60 (1.63) | 7.60 (1.41)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Improved Pain Relief and/or Convenience During the AdaptiveStim Programming Arm Relative to the Manual Programming Arm
Description: After subjects experienced both AdaptiveStim and manual programming at 16 weeks post-implant, subjects were asked to compare pain relief and convenience when they had AdaptiveStim ON to AdaptiveStim OFF in two separate domains using two 5-point Likert scales. The outcome measure for the primary objective is the percentage of subjects who report improved pain relief with no loss of convenience or improved convenience with no loss of pain relief during the AdaptiveStim programming arm relative to the manual programming arm. These subjects were considered successful for the primary objective.
Time Frame: 16 weeks post-implant
Population: The ITT analysis included 74 subjects; 2 randomized subjects, who discontinued early due to infections, were excluded per protocol. The 3 other subjects who discontinued early were included in ITT analysis and imputed as failures for the primary objective.
  No imputation method was used for 71 subjects included in the completed case analysis.
Measure: Number; unit: percentage of participants
Arm/Group | 6-week AdaptiveStim Followed by 6-week Manual Programming | 6-week Manual Followed by 6-week AdaptiveStim Programming
Number analyzed (Participants) | 34 | 40
percentage of participants
  Intent-to-treat analysis (n = 34, 40) | 91.2 | 82.5
  Completed case analysis (n = 33, 38) | 93.9 | 86.8
Statistical Analysis 1: Comparison: 6-week AdaptiveStim Followed by 6-week Manual Programming vs 6-week Manual Followed by 6-week AdaptiveStim Programming; ITT analysis: Hypothesis: The percentage of subjects who succeed must be greater than 25%. H0: p ≤ 0.25 HA: p > 0.25; Test type: Superiority or Other; p < 0.001, Fisher Exact; binomial proportion = 0.865, 97.5% CI 1-sided [lower limit 0.765] — In this ITT analysis, the combined percentage of subjects with improved pain relief and/or convenience during the AdaptiveStim programming relative to the manual programming in both groups was reported
Statistical Analysis 2: Comparison: 6-week AdaptiveStim Followed by 6-week Manual Programming vs 6-week Manual Followed by 6-week AdaptiveStim Programming; Completed case analysis; Test type: Superiority or Other; p < 0.001, Fisher Exact; binomial proportion = 0.901, 97.5% CI 1-sided [lower limit 0.807] — In this completed case analysis, the combined percentage of subjects with improved pain relief and/or convenience during the AdaptiveStim programming relative to the manual programming in both groups was reported

2. Secondary Outcome: Percentage of Subjects With Worsened Pain Relief When Using AdaptiveStim Compared to Manual Programming
Description: The pain relief question was a 5-point Likert scale question comparing pain relief when using AdaptiveStim programming relative to manual programming after subjects finished both programming periods. The choices were much worse pain relief with AdaptiveStim, somewhat worse pain relief with AdaptiveStim, no difference in pain relief, somewhat better pain relief with AdaptiveStim, and much better pain relief with AdaptiveStim. Subjects who had worsening pain relief were defined as subjects who responded "much worse pain relief with AdaptiveStim" or "somewhat worse pain relief with AdaptiveStim".
Time Frame: 16 weeks post-implant
Population: A total of 71 subjects with completed data were included in this analysis.
Measure: Number; unit: percentage of participants
Groups:
- 6-week Manual Followed by 6-week AdaptiveStime Programming: Subjects received manual programming for 6 weeks, followed by AdaptiveStim programming for 6 weeks.
Arm/Group | 6-week AdaptiveStim Followed by 6-week Manual Programming | 6-week Manual Followed by 6-week AdaptiveStime Programming
Number analyzed (Participants) | 33 | 38
percentage of participants | 0 [0.3% to 9.8%] | 5.3
Statistical Analysis 1: Comparison: 6-week AdaptiveStim Followed by 6-week Manual Programming vs 6-week Manual Followed by 6-week AdaptiveStime Programming; Test type: Superiority or Other; binomial proportion = 0.028, 95% CI 2-sided [0.003 to 0.098] — The combined percentage of subjects with worsened pain relief was reported

3. Secondary Outcome: Manual Adjustments Presented as Button Presses
Description: The number of individual adjustments, ie, button presses, were recorded automatically in the patient programmer, which was specifically designed for this study. The number of button presses per day for manual patient programmer adjustments during the manual programming arm and the AdaptiveStim programming arm of the study were compared.
Time Frame: Baseline, 10 weeks and 16 weeks post-implant
Population: Subjects with manual adjustments data from patient programmer were included in the analysis.
Measure: Mean (Standard Deviation); unit: Button presses per day
Groups:
- AdaptiveStim Treatment Arm: Subjects in AdaptiveStim treatment arm received programming provided by the RestoreSensor neurostimulator with AdaptiveStim ON.
- Manual Treatment Arm: Subjects in manual treatment arm received programming provided by the RestoreSensor neurostimulator with AdaptiveStim OFF.
Arm/Group | AdaptiveStim Treatment Arm | Manual Treatment Arm
Number analyzed (Participants) | 69 | 69
Button presses per day | 20.9 (41.4) | 35.7 (71.8)
Statistical Analysis 1: Comparison: AdaptiveStim Treatment Arm vs Manual Treatment Arm; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test; Mean Difference (Final Values) = 14.8, Standard Deviation 51.9

4. Secondary Outcome: NPRS Scores From Baseline to Follow-up Visits at 10 Weeks and 16 Weeks Post-implant
Description: The 11-point (ie, 0-10) numeric rating scale of pain intensity (NPRS) was used to assess the overall pain at baseline and follow-up visits. In the pain diary, subjects were presented a numeric scale with numbers from 0 to 10, with 0 meaning "No pain" and 10 meaning "Pain as bad as you can imagine," accompanied by the instructions "Please rate your pain by indicating the number that best describes your pain on average in the last 24 hours." The subjects were asked to complete a diary for 7 consecutive days before implant, 10 weeks, and 16 weeks post-implant visits.
Time Frame: Baseline, 10 weeks and 16 weeks post-implant
Population: 69 of the 76 subjects completed pain diary for both baseline and 10 weeks. 69 of the 76 subjects completed pain diary for both baseline and 16 weeks. Since 2 datasets had 2 different pairs of data due to different subjects who completed the pain diary, baseline NPRS in two analyses varied slightly.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- NPRS at Baseline (Subject With Score at 10 Weeks Post-implant); NPRS at 10 Weeks Post-implant: Included subjects with NPRS scores from both baseline and 10 weeks post-implant
- NPRS at Baseline (Subject With Score at 16 Weeks Post-implant); NPRS at 16 Weeks Post-implant: Included subjects with NPRS scores from both baseline and 16 weeks post-implant
Arm/Group | NPRS at Baseline (Subject With Score at 10 Weeks Post-implant) | NPRS at 10 Weeks Post-implant | NPRS at Baseline (Subject With Score at 16 Weeks Post-implant) | NPRS at 16 Weeks Post-implant
Number analyzed (Participants) | 69 | 69 | 69 | 69
units on a scale | 5.99 (1.82) | 4.22 (2.05) | 5.90 (1.81) | 4.41 (2.18)
Statistical Analysis 1: Comparison: NPRS at Baseline (Subject With Score at 10 Weeks Post-implant) vs NPRS at 10 Weeks Post-implant; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test; Mean Difference (Final Values) = 1.77, Standard Deviation 1.93
Statistical Analysis 2: Comparison: NPRS at Baseline (Subject With Score at 16 Weeks Post-implant) vs NPRS at 16 Weeks Post-implant; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test; Mean Difference (Final Values) = 1.50, Standard Deviation 2.04

ADVERSE EVENTS:
Time Frame: The time frame for safety reporting was from study enrollment to final visit. After implant, subjects were followed for an average duration of 16 weeks during which they experienced both manual and AdaptiveStim programming of the RestoreSensor device.
Groups:
- Overall Adverse Events: Overall adverse events were reported.
Arm/Group | Overall Adverse Events
Serious Adverse Events (participants affected / at risk) | 8/76
Other Adverse Events (participants affected / at risk) | 53/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Adverse Events (N=76)
Gastroenteritis (Infections and infestations) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Adverse Events (N=76)
Undesirable change in stimulation (General disorders) | 21 (25)
Change in sensation of stimulation (General disorders) | 4 (5)
Nasopharyngitis (Infections and infestations) | 7 (7)
Influenza (Infections and infestations) | 4 (4)
Depression (Psychiatric disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 4 (4)
Paraesthesia (Nervous system disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (17)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain (General disorders) | 9 (10)
Implant site irritation (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days